CLINICAL TRIAL: NCT06434844
Title: Effectiveness of Auricular Acupuncture in Reducing Dental Anxiety and Pain Perception During Orthodontic Extractions Among Adolescents - A Crossover Double-Blinded Randomised Controlled Trial
Brief Title: Effectiveness of Auricular Acupuncture in Reducing Dental Anxiety and Pain Perception During Orthodontic Extractions Among Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UW23-024
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; dental pain; auricular acupunctures
MeSH Terms: conditions — Toothache | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both acupuncture interventions will be carried out by a Hong Kong licenced Chinese medical practitioner (CMP) with no involvement in data collection and assessment. A research assistant will be responsible for the randomisation and inform the CMP regarding the group allocation. The acupuncture needles are kept in place for 20 minutes before the dental treatment.
  The extractions of premolars will be performed by a licenced general dental practitioner who is blinded towards the types of acupuncture received, so as the patient and their parents or caretakers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st visit Auricular acupuncture; 2nd visit Placebo sham acupuncture (Experimental): The subjects will receive auricular acupuncture in the 1st visit and placebo sham acupuncture in the 2nd visit.
  Interventions: Procedure: Auricular acupunctures; Procedure: Sham acupunctures
- 1st visit Placebo sham acupuncture; 2nd visit Auricular acupuncture (Sham Comparator): The subjects will receive placebo sham acupuncture in the 1st visit and auricular acupuncture in the 2nd visit.
  Interventions: Procedure: Auricular acupunctures; Procedure: Sham acupunctures

INTERVENTIONS:
Procedure: Auricular acupunctures — After disinfection of the external ear with 75% alcohol wipes, 018x 13 filiform needles (Mocm International Limited) will be used to perform the auricular acupunctures at the relaxation point, tranquilizer point and master cerebral point at the left and right external ears.
Procedure: Sham acupunctures — The auricular acupoints of finger, shoulder and tonsil will be targeted instead. These points are also located at the external ear and comparable to those in the intervention group. The external ear will be disinfected with 75% alcohol wipes. Auricular acupunctures with 018x 13 filiform needles (Mocm International Limited) will be carried out at the finger point, shoulder point and tonsil point of the left and right external ears.

SUMMARY:
This prospective, randomised, double-blinded cross-over study aims to compare the effectiveness of auricular acupuncture (AA) with placebo sham acupuncture (PSA) in reducing dental anxiety, pain perception and physiological responses to stress and anxiety among adolescents during orthodontic extractions.

Adolescents aged between 10-19 years old who are undergoing orthodontic treatments requiring bilateral premolar extractions will be invited to complete a validated questionnaire to record their dental anxiety level, oral health knowledge, attitudes, practices, demographic and socio-economic factors. During orthodontic extractions, physiological responses including heart rate and oxygen saturation will be measured with a fingertip pulse oximeter throughout the process.

The participants will be allocated randomly to one of the two groups in the study.

Group 1-- auricular acupuncture in their first orthodontic extraction visit and placebo sham acupuncture in their second orthodontic extraction visit.

Group 2-placebo sham acupuncture in their first orthodontic extraction visit and auricular acupuncture their second orthodontic extraction visit.

Both acupuncture interventions will be carried out by a Hong Kong registered Chinese medical practitioner. The acupuncture needles are kept in place for 20 minutes to exert its effect before the dental extraction. Placebo sham acupuncture will not cause any harm, but the acupuncture points have no reported effect on stress relief.

The extraction of premolars will be performed by a Hong Kong registered dentist. Local anesthesia is injected to numb the respective site, then the premolar will be removed with forceps, followed by stopping the bleeding by biting firmly on gauze.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthodontic treatment and require bilateral extraction of premolars.
* Have parental consent signed by their parent or guardian.
* Medically fit with either ASA I or II status
* Have not taken any medications, especially anxiolytics and antidepressants
* The premolars to be extracted should be fully erupted and without any signs of ankylosis.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental fear | Baseline, immediately after the intervention. immediately after the surgery
  Self-reported dental fear measured by Spielberger State Trait Anxiety Inventory score, Scores range from 20 to 80, with higher scores correlating with greater anxiety

SECONDARY OUTCOMES:
Pain perceived | Immediately after the intervention. immediately after the surgery
  Pain measured by Visual Analog Scale. Scores range from 0-10, with her scores correlating with greater pain
Psychological changes | Baseline, perioperatively, immediately after the surgery
  Heart rate
Psychological changes | Baseline, perioperatively, immediately after the surgery
  Saturation of peripheral oxygen (SpO2) measurement

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hksar PRC, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) and other supporting materials will be made available to other researchers upon valid requests to the PI of the study.